CLINICAL TRIAL: NCT03783325
Title: Assessing Gene-Environment Interactions in Clinical Presentation of Nevi and Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-1603.cc
Record Dates: First submitted 2018-12-13; First posted 2018-12-21 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Nevi and Melanomas
Keywords: Sun Exposure; UV Dosimetry; Biomarkers; Behaviors; Genetics
MeSH Terms: conditions — Nevi and Melanomas; Behavior

STUDY DESIGN:
Intervention Model Description: Patients will have the opportunity to participate in a questionnaire and then they are given the option to participate in substudy A (wear a UV dosimeter, complete questionnaires, and receive feedback based on the UV dosimeter results), subtstudy B (wear a skin patch, participate in a UV photo analysis, answer questionnaires), and/or substudy C (give biological samples via nevi).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UV Counseling (Other): Evaluate the effectiveness of dosimetry feedback on sun exposure behaviors, attitudes, and awareness in patients diagnosed with melanoma.
  Interventions: Behavioral: UV Counseling
- Visual Analysis - UV Photo (Experimental): Assess the relationships between UV camera score, silicone mold of a skin patch, phenotypic evaluation and sun-exposure behaviors. Technically, this arm is a sub-study that does not involve an intervention. Patients are not receiving an intervention; they are simply providing data to the study team.
  Interventions: Other: UV Photo
- Biological Sample (Experimental): Determine the relationship between measures of sun exposure and genomic characteristics of tumors in melanoma patients. Technically, this arm is a sub-study that does not involve an intervention. Patients are not receiving an intervention; they are simply providing data to the study team.
  Interventions: Other: Biological Sample

INTERVENTIONS:
Behavioral: UV Counseling — This is a sub-study that involves a behavioral intervention. Participants will wear a UV dosimetry for 3 weeks, return the device and receive feedback. After the feedback, they will re-wear the device for an additional 3 weeks.
  Arms: UV Counseling
Other: UV Photo — Technically, this arm is a sub-study that does not involve an intervention. Patients are not receiving an intervention; they are simply providing data to the study team.
  Arms: Visual Analysis - UV Photo
Other: Biological Sample — Technically, this arm is a sub-study that does not involve an intervention. Patients are not receiving an intervention; they are simply providing data to the study team.
  Arms: Biological Sample

SUMMARY:
This research study is designed to better understand the role of genetics, sun-exposure and phenotypic factors in melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. > or = 18 years of age
2. Patient at the University of Colorado Anschutz Medical Campus Cutaneous Oncology Clinic or Dermatology Clinic OR attend the fundraising event of the Colorado Melanoma Foundation

Exclusion Criteria:

1. No exclusion criteria listed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Sun Exposure Behaviors | Start of study, initial interaction with participants.
  A short questionnaire is administered during the clinic visit to assess sun exposure behaviors of melanoma patients. The data gathered from this questionnaire will help identify possible trends in sun exposure behaviors and provide a baseline dataset for future research,
UV Exposure Assessment | Start of study to end of study, up to 6 weeks
  Identify the difference between self-reported sun exposure behavior and actual UV exposure by having patients wear individual dosimeters
Visual Appearance Relationships: Melanoma, Questionnaire | Start of study to end of study, up to 3 years
  Determine the relationship between UV camera score, skin patch, sun exposure history, and phenotypic evaluation in melanoma patients using a sun exposure questionnaire
Visual Appearance Relationships: Non-Melanoma , Questionnaire | Start of study to end of study, up to 3 years
  Determine the relationship between UV camera score, skin patch, sun exposure history, and phenotypic evaluation in non-melanoma patients using a sun exposure questionnaire
Visual Appearance Relationships: Melanoma, Photography | Start of study to end of study, up to 3 years
  Determine the relationship between UV camera score, skin patch, sun exposure history, and phenotypic evaluation in melanoma patients using a UV photography
Visual Appearance Relationships: Non-Melanoma, Photography | Start of study to end of study, up to 3 years
  Determine the relationship between UV camera score, skin patch, sun exposure history, and phenotypic evaluation in non-melanoma patients using a UV photography
Visual Appearance Relationships: Melanoma, Casting | Start of study to end of study, up to 3 years
  Determine the relationship between UV camera score, skin patch, sun exposure history, and phenotypic evaluation in melanoma patients using a silicone casts
Visual Appearance Relationships: Non-Melanoma, Casting | Start of study to end of study, up to 3 years
  Determine the relationship between UV camera score, skin patch, sun exposure history, and phenotypic evaluation in non-melanoma patients using a silicone casts
Visual Appearance Relationships: Melanoma, SCINEXA | Start of study to end of study, up to 3 years
  Determine the relationship between UV camera score, skin patch, sun exposure history, and phenotypic evaluation in melanoma patients using a SCINEXA exam.
Visual Appearance Relationships: Non-Melanoma, SCINEXA | Start of study to end of study, up to 3 years
  Determine the relationship between UV camera score, skin patch, sun exposure history, and phenotypic evaluation in non-melanoma patients using a SCINEXA exam.
Genetics Correlations | Start of study to end of study, up to 3 years
  Determine whether UV exposure and camera scores correlates with UV signature (somatic) mutations and other tumor-related mutations in clinically benign nevi and primary melanomas using saliva samples, benign nevi, and primary melanomas. Next Generation Sequencing (NGS) will be used to obtain the genetic information from all samples.

SECONDARY OUTCOMES:
Self Reporting Behaviors | Start of study to end of study, up to 3 years
  Determine self-reported sun exposure behaviors through participant interviews. Questions are related to time spent outside, and what attempts to be sun-safe occurred while outside.
Behavioral Intervention and Immediate Follow Up | After wearing dosimetry for 3 weeks
  Participants will receive a personalized feedback plan and the success of the plan will be measured through individual dosimetry. We will track real time change in sun exposure based on repeat UV dosimetry.
Benign Nevi, DNA | Start of study to end of study, up to 3 years
  Determine if a relationship exists between the phenotypic attributes of benign nevi through analysis of genomic DNA
Benign Nevi, Mutations | Start of study to end of study, up to 3 years
  Determine if a relationship exists between the phenotypic attributes of benign nevi through analysis of somatic mutations
Benign Nevi, Exposure | Start of study to end of study, up to 3 years
  Determine if a relationship exists between the phenotypic attributes of benign nevi through analysis of analysis of UV exposure history
Benign Nevi, UV Camera | Start of study to end of study, up to 3 years
  Determine if a relationship exists between the phenotypic attributes of benign nevi through analysis of analysis of UV camera scores with the clinical presentation
Primary Melanomas, DNA | Start of study to end of study, up to 3 years
  Determine if a relationship exists between the phenotypic attributes of primary melanomas through analysis of genomic DNA
Primary Melanomas, Mutations | Start of study to end of study, up to 3 years
  Determine if a relationship exists between the phenotypic attributes of primary melanomas through analysis of somatic mutations
Primary Melanomas, Exposure | Start of study to end of study, up to 3 years
  Determine if a relationship exists between the phenotypic attributes of primary melanomas through analysis of UV exposure history
Primary Melanomas, UV Camera | Start of study to end of study, up to 3 years
  Determine if a relationship exists between the phenotypic attributes of primary melanomas through analysis of UV camera scores with the clinical presentation

CONTACTS AND LOCATIONS:
Overall Officials: Neil Box, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States